CLINICAL TRIAL: NCT03601559
Title: The Cognitive Effects of 6 Weeks Administration With a Probiotic: a Randomized, Placebo Controlled Proof-of-concept Study in Healthy Elderly Humans
Brief Title: The Cognitive Effects of 6 Weeks Administration With a Probiotic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: DuPont Nutrition and Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: NH-03937
Record Dates: First submitted 2018-07-05; First posted 2018-07-26 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2018-09

CONDITIONS: Cognitive Change
Keywords: gut-brain axis, cognitve demand battery, probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus paracasei Lpc-37 (Active Comparator): Probiotic
  Interventions: Dietary Supplement: Lactobacillus paracasei Lpc-37
- Placebo (Placebo Comparator): Inert placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus paracasei Lpc-37 — Live probiotic bacteria
  Arms: Lactobacillus paracasei Lpc-37
Dietary Supplement: Placebo — Inert placebo matched for taste and appearance
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the cognitive and mood effects of a probiotic dietary supplement when taken daily for 42 days in healthy older adults aged 65+

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥ 65 years
2. Willing and able to provide written and informed consent
3. Ability of the participant (in the Principal Investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects
4. Agreement to comply with the protocol and study restrictions
5. Available for all study visits
6. In good general health, self-reported and as judged by the Principal Investigator/Clinical advisor based on medical history
7. Fluent in written and spoken English
8. Participant is willing to maintain habitual diet (including caffeine and alcohol) and physical activity patterns throughout the study period
9. Has a bank account (required for payment)

Exclusion criteria:

1. Have any pre-existing significant acute or chronic co-existing medical condition / illness which contraindicates, in the Principal Investigator's judgement, entry to the study NOTE: the explicit exceptions to this are controlled (medicated) hypertension, arthritis, asthma, hay fever, high cholesterol and reflux-related conditions. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progess to screening if they have a condition/illness which would not interact with the active treatments or impede performance
2. History of dementia, stroke and other neurological conditions
3. Traumatic loss of consciousness in the last 12 months
4. History of epilepsy or Parkinson's disease
5. Anxiety, depression or any psychiatric disorder that the Principal Investigator believes would interfere with the objectives of the study and requiring treatment in the last 2 years
6. Currently taking (from day of screening onwards) or have previously taken (last 4 weeks prior to screening) prescription medications that the Principal Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results such as psychoactive medication (anxiolytics, sedatives, hypnotics, anti-psychotics, anti-depressants, anti-convulsants, centrally acting corticosteroids, opioid pain relievers) NOTE: the explicit exceptions to this are hormone replacement treatments for female participants where symptoms are stable, those medications used in the treatment of arthritis, high blood pressure, high cholesterol and reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, participants may be able to progress to screening
7. Currently taking (from day of screening onwards) medication or dietary supplements that the Principal Investigator believes would interfere with the objectives of the study, pose a safety risk or confound the interpretation of the study results such as: melatonin, vitamin E, multivitamins, B vitamin complex, ginkgo biloba, fish oil, St. John's Wort or other cognitive enhancing dietary or herbal supplements over the study period
8. Recent (within last 4 weeks prior to screening) or ongoing antibiotic therapy during the intervention period
9. Daily consumption of concentrated sources of probiotics and / or prebiotics within 2 weeks of screening and throughout the intervention period other than the provided study products (e.g., probiotic / prebiotic tablets, capsules, drops or powders), including yoghurt or yoghurt drinks
10. Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
11. Have a Body Mass Index (BMI) outside of the range 18.5-29.9 kg/m2
12. Have learning difficulties, dyslexia
13. Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
14. Current smoker (use of nicotine replacement products, vaping, gum, patches etc)
15. Have a history of alcohol or drug abuse
16. Current misuse of alcohol, drug or prescription medications
17. Excessive caffeine intake (>500 mg per day)
18. Excessive alcohol consumption (drinking on 5 or more days a week or consuming > 6 units of alcohol in a single session on 5 or more days a week) for 3 weeks prior to screening and during the intervention period
19. Contraindication to any substance in the investigational product
20. Principal Investigator believes that the participant may be uncooperative and / or noncompliant and should therefore not participate in the study
21. Participant under legal or administrative supervision
22. Have food intolerances / sensitivities
23. Have any health condition that would prevent fulfilment of the study requirements
24. Are unable or unwilling to complete all the study assessments
25. Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Episodic memory score | 6 weeks
  This is a composite measure derived from summing the z score performance on the following cognitive tasks: immediate word recall, delayed word recall, delayed picture recognition, delayed word recognition (-4 to 4)

SECONDARY OUTCOMES:
STAI-state total score | 6 weeks
  State-trait anxiety inventory 'state' total score (20-80)
STAI-trait total score | 6 weeks
  State-trait anxiety inventory 'trait' total score (20-80)
Accuracy of attention score | 6 weeks
  This is a composite measure derived from summing the z score accuracy performance on the choice reaction time and Rapid visual information processing tasks (-2 to 2)
Speed of attention score | 6 weeks
  This is a composite measure derived from summing the z score reaction times from the choice reaction time and Rapid visual information processing task (-2 to 2)
Working memory score | 6 weeks
  This is a composite measure derived from summing the z score accuracy performance on the numeric working memory task and Corsi block-tapping task (-2 to 2)
Speed of memory score | 6 weeks
  This is a composite measure derived from summing the z score reaction times on the numeric working memory task, the delayed name / face recall task, the delayed picture recognition task and the delayed word recognition task (-4 to 4)
Delayed word recall correct | 6 weeks
  total number of correctly identified words (0-15)
Delayed word recall errors | 6 weeks
  total number of error responses
Picture recognition reaction time | 6 weeks
  (ms)
Picture recognition accuracy | 6 weeks
Word recognition reaction time | 6 weeks
  (ms)
Word recognition accuracy | 6 weeks
Name to Face Recall correct responses | 6 weeks
  number
Name to Face Recall reaction time | 6 weeks
  (ms)
Peg and Ball task Planning time | 6 weeks
  (ms)
Peg and Ball task Completion time | 6 weeks
  (ms)
Peg and Ball task errors | 6 weeks
  Number
Stroop task accuracy | 6 weeks
Stroop task reaction time | 6 weeks
  (ms)
Immediate word recall task correctly identified words | 6 weeks
  total number (0-15)
Immediate word recall task error responses | 6 weeks
  total number
Numeric working memory accuracy | 6 weeks
Numeric working memory reaction time | 6 weeks
  (ms)
Choice reaction time accuracy | 6 weeks
Choice reaction time reaction time | 6 weeks
  (ms)
Rapid visual information processing accuracy | 6 weeks
Rapid visual information processing reaction time | 6 weeks
  (ms)
Rapid visual information processing false alarms | 6 weeks
  number
Corsi blocks accuracy | 6 weeks
  Average scores from the last five correctly completed trials from the Corsi block-tapping task
Rapid visual information processing accuracy | 6 weeks
  (%) - calculated from the 3 cycles of the Cognitive Demand Battery
Rapid visual information processing reaction time | 6 weeks
  (ms) - calculated from the 3 cycles of the Cognitive Demand Battery
Rapid visual information processing false alarms | 6 weeks
  number - calculated from the 3 cycles of the Cognitive Demand Battery
Serial 3 subtractions total responses | 6 weeks
  number- calculated from the 3 cycles of the Cognitive Demand Battery
Serial 3 subtractions total error responses | 6 weeks
  number - calculated from the 3 cycles of the Cognitive Demand Battery
Serial 7 subtractions total responses | 6 weeks
  number - calculated from the 3 cycles of the Cognitive Demand Battery
Serial 7 subtractions total error responses | 6 weeks
  number - calculated from the 3 cycles of the Cognitive Demand Battery
Mental fatigue | 6 weeks
  visual analogue scale (%) - calculated from the 3 cycles of the Cognitive Demand Battery
Alertness | 6 weeks
  visual analogue scale (%) - calculated from the 3 cycles of the Cognitive Demand Battery
Alert | 6 weeks
  derived from Bond Lader visual analogue scale
Content | 6 weeks
  derived from Bond Lader visual analogue scale
Calm | 6 weeks
  derived from Bond Lader visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Philippa A Jackson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study site website — http://nutrition-neuroscience.co.uk